CLINICAL TRIAL: NCT03232684
Title: Rapid On-site Evaluation of EBUS-TBNA Samples From Intrathoracic Lymphadenopathy; Can it be Reliably Performed by a Pulmonologist?
Brief Title: Rapid On-site Evaluation of Endobronchial Ultrasound Guided Transbronchial Needle Aspiration Samples by Pulmonologists
Status: Completed | Type: Observational
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Principal Investigator, Rocco Trisolini, Director, Interventional Pulmonology Unit, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: CE 17021
Record Dates: First submitted 2017-07-21; First posted 2017-07-28 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Intrathoracic Lymphadenopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid on-site evaluation — On-site (endoscopy suite) evaluation, by a pathologist or a pulmonologist, of specimens retrieved from intrathoracic lymph nodes during EBUS-TBNA

SUMMARY:
The study is aimed at verifying if a pulmonologist in training can reliably assess the adequacy of EBUS-TBNA samples from intrathoracic lymphadenopathy after a period of training provided by an experienced pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Indication to sampling of intrathoracic lymphadenopathy based on computed tomography (CT) and/or positron emission tomography (PET)/CT findings
* Signed informed consent

Exclusion Criteria:

* High risk conditions for the performance of bronchoscopy and endobronchial ultrasound guided transbronchial needle aspiration (EBUS-TBNA)
* High risk condition for deep sedation (ASA 4)
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with enlarged intratoracic lymph nodes
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Accuracy with which the pulmonologist will identify inadequate EBUS-TBNA samples | Up to 1 week
  The Outcome 1 will be measured by verifying the agreement between the pulmonologist judgment and the pathologist judgment, the latter being the gold standard

SECONDARY OUTCOMES:
Accuracy with which the pulmonologist will be able, in case of adequate EBUS-TBNA sample, to assign the specimen to one of the following specific diagnoses: 1) reactive lymph node; 2) malignancy; 3) granulomatous inflammation | Up to 1 week
  The Outcome 1 will be measured by verifying the agreement between the pulmonologist judgment and the pathologist judgment, the latter being the gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Policlinico S. Orsola & Maggiore Hospitals
Locations (1):
- Maggiore Hospital, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trisolini R, Cancellieri A, Tinelli C, Paioli D, Scudeller L, Casadei GP, Forti Parri S, Livi V, Bondi A, Boaron M, Patelli M. Rapid on-site evaluation of transbronchial aspirates in the diagnosis of hilar and mediastinal adenopathy: a randomized trial. Chest. 2011 Feb;139(2):395-401. doi: 10.1378/chest.10-1521. Epub 2010 Oct 28. PMID 21030491
- [Result] Bonifazi M, Sediari M, Ferretti M, Poidomani G, Tramacere I, Mei F, Zuccatosta L, Gasparini S. The role of the pulmonologist in rapid on-site cytologic evaluation of transbronchial needle aspiration: a prospective study. Chest. 2014 Jan;145(1):60-65. doi: 10.1378/chest.13-0756. PMID 23846345